CLINICAL TRIAL: NCT04860999
Title: The Ability of Osteopathic Structural Evaluation to Assess Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-051
Record Dates: First submitted 2021-03-24; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Osteopathic Manipulation; Postural; Defect; Somatic; Functional Disturbance
Keywords: gait; assessment; manipulation; asymmetry; osteopathic
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Participants underwent an osteopathic structural examination and osteopathic manipulation. Participants completed a biomechanical assessment prior to and following the osteopathic manipulation to evaluate the effect of osteopathic manipulation on gait asymmetry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Somatic Dysfunction (Experimental): This is the single study arm. All participants completed an osteopathic postural examination and an osteopathic manipulative treatment. Participants also completed a biomechanical assessment prior to and following the osteopathic manipulative treatment to evaluate effects of the treatment on the gait asymmetry.
  Interventions: Procedure: Osteopathic Manipulative Treatment

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — The osteopathic manipulations focused on treating the asymmetric postural dysfunction that was identified by the initial functional structural evaluation. The manipulation consisted of typical time-honored osteopathic treatments directed at the identified somatic dysfunction(s). These techniques were clinically directed and include: soft tissue, muscle energy, high velocity low amplitude, low velocity high amplitude as well as facilitated positional release as indicated.

SUMMARY:
Movement and loading asymmetry have been associated with injury risk for a variety of both acute and chronic musculoskeletal injuries. In addition, asymmetric movements have been identified as compensatory strategies to allow for ambulation in a variety of post-operative populations. Osteopathic physicians have been assessing both structure and function through the use of structural evaluation techniques along with postural assessment that can identify somatic dysfunction. However, no studies have identified the ability of an osteopathic structural evaluation and postural assessment to identify potential movement disorders and loading asymmetry. Therefore, the primary objective of this study is to determine the acute impact of an osteopathic manipulation on restoration of side-to-side symmetry during walking gait in participants who are categorized as having lower extremity dysfunction. We enrolled 51 participants who are pain-free and without a history of major orthopaedic injuries that required surgical intervention. Each subject completed an osteopathic structural evaluation and postural assessment along with an osteopathic manipulation. All participants completed instrumented gait analyses before and after the osteopathic manipulation using a motion capture system and an instrumented treadmill to determine the participant's movement and loading asymmetry during walking.

DETAILED DESCRIPTION:
Following recruitment and the completion of informed consent, each subject had a standard osteopathic postural assessment. This assessment was completed by a single experienced osteopathic physicians who uses manual medicine techniques in clinical practice as well as teaching these techniques to osteopathic medical students.

Following the osteopathic exam, all participants completed an initial biomechanical assessment in the Kevin P. Granata Biomechanics Lab at Virginia Tech. All subjects wore form fitting shorts and a shirt, plus a pair of athletic shoes (Nike Pegasus, Nike Inc, Beaverton, CO) all of which was provided for them to use during testing. Patients had retro-reflective markers attached at specific locations on both lower extremities to track segmental motion level walking. Three-dimensional coordinate data was collected using a 8-camera motion capture system at a sampling rate of 120 Hz (Qualysis, Sweden). Ground reaction forces were collected using an instrumented treadmill with a sampling rate of 1440 Hz (AMTI, Watertown, Massachusetts). Each subject completed a standing trial followed by 2 walking trials. Participants completed 5 minutes of continuous steady state walking at 1.5m/s on the instrumented treadmill. Participants then completed a second 5 minute walking trial at their self-selected speed on the instrumented treadmill. During both 5 minute walking trials, data was collected simultaneously from the motion capture system and the instrumented treadmill from minute 1 through minute 4 in order to avoid collection during the beginning and end of the trial.

After the initial biomechanical examination, osteopathic manipulation was performed on participants in the Dysfunction group. The osteopathic manipulations were focused on treating the asymmetric postural dysfunction that was identified by the initial functional structural evaluation. The manipulation consisted of typical time-honored osteopathic treatments directed at the identified somatic dysfunction(s). These techniques were clinically directed and include: soft tissue, muscle energy, high velocity low amplitude, low velocity high amplitude as well as facilitated positional release as indicated.

After the osteopathic manipulation, participants completed the same walking assessment for a second time. This immediate post-biofeedback testing was completed using the same protocol as the baseline assessment previously described.

All osteopathic assessments and manipulations were completed by a single experienced osteopathic clinicians and the biomechanical assessments was completed by a second individual using a standard set of directions.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 and 35

Exclusion Criteria:

* History of major lower extremity surgery
* Currently being under the care of a medical professional for any musculoskeletal injury or chronic condition

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Peak vertical ground reaction force asymmetry between limbs during the weight acceptance and propulsive phases of walking | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Peak vertical ground reaction force asymmetry between limbs during the weight acceptance and propulsive phases of walking | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)

SECONDARY OUTCOMES:
Peak vertical ground reaction force impulse asymmetry between limbs | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Peak knee flexion angle asymmetry between limbs | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Step length asymmetry between limbs | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Stride length asymmetry between limbs | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Stance time asymmetry between limbs | Before an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5-10 minutes before)
Peak vertical ground reaction force impulse asymmetry between limbs | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)
Peak knee flexion angle asymmetry between limbs | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)
Step length asymmetry between limbs | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)
Stride length asymmetry between limbs | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)
Stance time asymmetry between limbs | After an osteopathic manipulative treatment addressing identified somatic dysfunctions (approximately 5 minutes after)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Queen, Principal Investigator — Virginia Polytechnic Institute and State University; Gunnar Brolinson, Principal Investigator — Edward Via College of Osteopathic Medicine; Mark Rogers, Principal Investigator — Edward Via College of Osteopathic Medicine
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No